CLINICAL TRIAL: NCT00402324
Title: A Double-Blind Placebo Controlled Trial of Divalproex and Olanzapine in Bipolar I Disorder, Mixed Episode
Brief Title: A Comparison of Olanzapine in Combination With a Mood Stabilizer vs Mood Stabilizer Alone, in Mixed Bipolar Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 10825; F1D-US-HGMO
Record Dates: First submitted 2006-11-17; First posted 2006-11-22 (Estimated); Results first posted 2009-05-27 (Estimated); Last update posted 2009-06-03 (Estimated); Status verified 2009-05

CONDITIONS: Bipolar I Disorder
Keywords: Mixed episode associated with Bipolar I
MeSH Terms: interventions — Olanzapine; Valproic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Experimental): olanzapine and divalproex
  Interventions: Drug: olanzapine; Drug: divalproex
- 2 (Placebo Comparator): placebo and divalproex
  Interventions: Drug: placebo; Drug: divalproex

INTERVENTIONS:
Drug: olanzapine — 15mg, capsules, by mouth every evening, daily for minimum of one day, followed by 5-20mg, capsules, by mouth every evening, daily for remainder of study (6 weeks total).
  Other Names: LY170053; Zyprexa
  Arms: 1
Drug: placebo — placebo, capsules, by mouth every evening, daily, for 6 weeks.
  Arms: 2
Drug: divalproex — dose to maintain blood levels of 75-125 ug/mL, by mouth, twice a day, daily for 52 days (Study Period I and Study Period II).

SUMMARY:
Whether treatment with olanzapine in combination with mood stabilizer reduces symptoms of both mania and depression more than treatment with mood stabilizer alone, in patients with a mixed episode of bipolar I disorder.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with a mixed episode of bipolar I disorder.
* Have had at least one previous manic or mixed episode associated with bipolar disorder
* You must be between 18 and 60 years old.
* You must be able to visit the doctor's office three times in the first week and then once every week for the next five weeks.
* If you are a female, you must have a negative pregnancy test and be using an effective method of contraception.

Exclusion Criteria:

* You have a diagnosis of schizophrenia, schizoaffective disorder or substance abuse or dependence.
* You have diseases of the intestinal tract, lungs, liver, kidney, nervous or endocrine systems, or blood.
* Have required a recent thyroid hormone supplement to treat hypothyroidism (must have been on a stable dose of the medication for at least 2 months prior to Visit 3).
* You are allergic to any of the medications involved in this study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 202 (Actual)
Dates: Start 2006-12; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hialeah, Florida, United States

REFERENCES:
- [Derived] Houston JP, Gatz JL, Degenhardt EK, Jamal HH. Symptoms predicting remission after divalproex augmentation with olanzapine in partially nonresponsive patients experiencing mixed bipolar I episode: a post-hoc analysis of a randomized controlled study. BMC Res Notes. 2010 Nov 2;3:276. doi: 10.1186/1756-0500-3-276. PMID 21044339
- [Derived] Houston JP, Tohen M, Degenhardt EK, Jamal HH, Liu LL, Ketter TA. Olanzapine-divalproex combination versus divalproex monotherapy in the treatment of bipolar mixed episodes: a double-blind, placebo-controlled study. J Clin Psychiatry. 2009 Nov;70(11):1540-7. doi: 10.4088/JCP.08m04895yel. Epub 2009 Sep 22. PMID 19778495
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study Period 1 was a 2-28 day day period allowing for screening, divalproex treatment initiation (if appropriate) and washout. Patients meeting diagnostic criteria and having therapeutic serum levels of divalproex in target range of 75 to 125 µg/mL (≥80 µg/mL recommended) during Study Period I, will be randomized into either placebo or olanzapine.
Groups:
- Olanzapine: Olanzapine: 15mg, capsules, by mouth every evening, daily for minimum of one day, followed by 5-20mg, capsules, by mouth every evening, daily for remainder of study (6 weeks total).
  Divalproex: dose to maintain blood levels of 75-125 ug/mL, by mouth, twice a day, daily for 6 weeks (following dose achieved in Study Period I).
- Placebo: Placebo: placebo capsules, by mouth every evening, daily, for 6 weeks. Divalproex: dose to maintain blood levels of 75-125 ug/mL, by mouth, twice a day, daily for 6 weeks (following dose achieved in Study Period I).
Period: Overall Study
Arm/Group | Olanzapine | Placebo
Started | 101 | 101
Completed | 58 | 60
Not Completed | 43 | 41
Not completed — Lost to Follow-up | 11 | 11
Not completed — Protocol Entry Criteria Not Met | 5 | 4
Not completed — Protocol Violation | 8 | 7
Not completed — Withdrawal by Subject | 5 | 2
Not completed — Physician Decision | 2 | 4
Not completed — Sponsor Decision | 4 | 5
Not completed — Lack of Efficacy | 1 | 4
Not completed — Adverse Event | 6 | 4
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Olanzapine | Placebo | Total
Number analyzed (Participants) | 101 | 101 | 202
Age Continuous [Mean (Standard Deviation); unit: years] | 38.61 (11.20) | 38.52 (11.07) | 38.56 (11.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 58 | 119
  Male | 40 | 43 | 83
Region of Enrollment [Number; unit: participants]
  United States | 101 | 101 | 202
Race/Ethnicity [Number; unit: participants]
  Caucasian | 46 | 56 | 102
  African Descent | 38 | 29 | 67
  Hispanic | 15 | 13 | 28
  Native American | 1 | 2 | 3
  East Asian | 1 | 1 | 2
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms per square meters] — Body mass index is an estimate of body fat based on body weight divided by height squared.
  kilograms per square meters | 30.73 (8.99) | 31.72 (8.29) | 31.23 (8.64)
Body Weight [Mean (Standard Deviation); unit: kilograms] | 87.33 (24.17) | 90.75 (23.70) | 89.04 (23.94)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Young Mania Rating Scale (YMRS) Scores From Baseline to Endpoint.
Description: The YMRS is an 11-item scale that measures the severity of manic episodes. Four items are rated on a scale from 0 (symptom not present) to 8 (symptom extremely severe). The remaining items are rated on a scale from 0 (symptom not present) to 4 (symptom extremely severe). The YMRS total score ranges from 0 to 60.
Time Frame: Baseline to endpoint (6 weeks)
Population: Intent to Treat analysis. All randomized patients with baseline & at least one post-baseline measure.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Olanzapine | Placebo
Number analyzed (Participants) | 100 | 101
units on a scale | -10.15 (0.44) | -7.68 (0.44)
Statistical Analysis 1: Comparison: Olanzapine vs Placebo; The overall power of the two co-primary analyses-the probability of simultaneously rejecting both co-primary null hypotheses-for this sample size under assumed effect sizes of 0.5 and 0.45 is estimated as approximately 85-87% and 77-80%, respectively; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — All tests of treatment effects will be conducted at a two-sided alpha level of 0.05 unless otherwise stated; Mixed Model Repeated Measures (MMRM) Change = Therapy PooledINV Visit Baseline Baseline*Visit Therapy*Visit. P-value from therapy term in model

2. Primary Outcome: Mean Change in Hamilton Depression Rating Scale-21 (HAMD) Scores From Baseline to Endpoint.
Description: The 21-item HAMD measures depression severity. Items are rated on a scale from 0 (symptoms not present) to a maximum of 2 to 4 (symptom extremely severe) for a total score range of 0 to 60.
Time Frame: Baseline to endpoint (6 weeks)
Population: Intent to Treat analysis. All randomized patients with baseline & at least one post-baseline measure.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Olanzapine | Placebo
Number analyzed (Participants) | 100 | 101
units on a scale | -9.37 (0.55) | -7.69 (0.54)
Statistical Analysis 1: Comparison: Olanzapine vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.022, Mixed Models Analysis — All tests of treatment effects will be conducted at a two-sided alpha level of 0.05 unless otherwise stated; [statistical method as in outcome 1, analysis 1]

3. Secondary Outcome: Number of Participants Meeting the Criteria for Mixed Onset of Action
Description: The original outcome measure was Time to Mixed Onset of Action (at least a 25% reduction on HAMD and YMRS total scores from baseline); however since upper limit of measure of dispersion could not be computed by observed data, which is not allowed on this system, number of patients with event are presented instead.
Time Frame: Baseline to endpoint (6 weeks)
Population: All randomized participants with both baseline and post-baseline measures. Intention to Treat analysis.
Measure: Number; unit: participants
Arm/Group | Olanzapine | Placebo
Number analyzed (Participants) | 100 | 101
participants | 81 [3 to 15] | 71 [4 to 45]
Statistical Analysis 1: Comparison: Olanzapine vs Placebo; Test type: Superiority or Other; p = 0.100, Fisher Exact

4. Secondary Outcome: Number of Participants Meeting the Criteria for Mixed Response
Description: The original outcome measure was Time to Mixed Response(at least a 50% reduction on HAMD and YMRS total scores from baseline); however since upper limit of measure of dispersion could not be computed by observed data, which is not allowed on this system, number of patients with event are presented instead.
Time Frame: baseline to endpoint (6 weeks)
Population: All randomized participants with both baseline and post-baseline measures. Intention to Treat analysis.
Measure: Number; unit: participants
Arm/Group | Olanzapine | Placebo
Number analyzed (Participants) | 100 | 101
participants | 54 [lower limit 9] | 40 [lower limit 13]
Statistical Analysis 1: Comparison: Olanzapine vs Placebo; Test type: Superiority or Other; p = 0.048, Fisher Exact

5. Secondary Outcome: Mean Change in Clinical Global Impression for Bipolar Illness Severity (CGI-BP) From Baseline to Endpoint
Description: CGI-BP Severity is used by the clinician to record the severity of illness at the time of assessment. The score ranges from 1 (normal, not at all ill) to 7 (among the most extremely ill patients).
Time Frame: Baseline to endpoint (6 weeks)
Population: Intent to Treat analysis. Number of randomized patients with baseline and at least one nonmissing postbaseline value. Last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Olanzapine | Placebo
Number analyzed (Participants) | 100 | 101
units on a scale | -1.34 (0.11) | -1.06 (0.11)
Statistical Analysis 1: Comparison: Olanzapine vs Placebo; Test type: Superiority or Other; p = 0.056, ANCOVA; Type III sums of squares of ANCOVA model: Change= TRT + Pooled Investigator + Baseline

6. Secondary Outcome: Number of Patients Hospitalized Due to Relapse of Mania or Depression.
Description: Number of participants hospitalized as a result of relapse of mania or depression.
Time Frame: Baseline to endpoint (6 weeks)
Population: Intent to Treat analysis. All randomized patients.
Measure: Number; unit: participants
Arm/Group | Olanzapine | Placebo
Number analyzed (Participants) | 101 | 101
participants | 1 | 0

7. Secondary Outcome: Clinically Significant Laboratory Values - Fasting Cholesterol Change From Baseline
Description: Change from Baseline to endpoint in cholesterol: value of cholesterol measure at endpoint minus the value at baseline.
Time Frame: Baseline to endpoint (6 weeks)
Population: All randomized participants with both baseline and at least one post-baseline measure. Intention to Treat analysis.
Measure: Mean (Standard Deviation); unit: milligrams per deciliter
Arm/Group | Olanzapine | Placebo
Number analyzed (Participants) | 62 | 68
milligrams per deciliter
  Total Cholesterol Baseline | 191.37 (41.23) | 192.25 (44.45)
  Total Cholesterol Change from Baseline | -7.80 (31.77) | -8.72 (28.80)
  Low Density Lipoprotein Baseline (N=62,N=64) | 115.32 (38.82) | 111.01 (36.74)
  Low Density Lipoprotein Change (N=62,N=64) | -9.22 (27.31) | -9.77 (28.05)
  High Density Lipoprotein Baseline | 53.76 (12.03) | 51.48 (11.64)
  High Density Lipoprotein Change from Baseline | -3.24 (10.02) | -1.22 (8.90)
Statistical Analysis 1: Comparison: Olanzapine vs Placebo; Test type: Superiority or Other; p = 0.657, ANOVA — P-value for Total Cholesterol Change from Baseline; Type III sums of squares of ANOVA model: Ranked Change= Treatment + Pooled Investigator
Statistical Analysis 2: Comparison: Olanzapine vs Placebo; Test type: Superiority or Other; p = 0.924, ANOVA — P-value for Low Density Lipoprotein Change from Baseline; Type III sums of squares of ANOVA model: Ranked Change= Treatment + Pooled Investigator
Statistical Analysis 3: Comparison: Olanzapine vs Placebo; Test type: Superiority or Other; p = 0.122, ANOVA — P-value for High Density Lipoprotein Change from Baseline; Type III sums of squares of ANOVA model: Ranked Change= Treatment + Pooled Investigator

8. Secondary Outcome: Clinically Significant Laboratory Values - Fasting Triglycerides Change From Baseline
Description: Change from baseline to endpoint in triglycerides: Value of triglyceride measure at endpoint minus value at baseline.
Time Frame: Baseline to endpoint (6 weeks)
Population: All randomized participants with both baseline and post-baseline measures. Intention to Treat analysis.
Measure: Mean (Standard Deviation); unit: milligrams per deciliter
Arm/Group | Olanzapine | Placebo
Number analyzed (Participants) | 62 | 68
milligrams per deciliter
  Baseline | 111.46 (61.54) | 139.75 (77.22)
  Change from Baseline | 22.91 (67.70) | 16.80 (73.25)
Statistical Analysis 1: Comparison: Olanzapine vs Placebo; Test type: Superiority or Other; p = 0.293, ANOVA — P-value for Fasting Triglycerides Change from Baseline; Type III sums of squares of ANOVA model: Ranked Change= Treatment + Pooled Investigator

9. Secondary Outcome: Clinically Significant Laboratory Values - Fasting Blood Glucose Change From Baseline
Description: Change from baseline to endpoint in fasting blood glucose: Value of fasting blood glucose measure at endpoint minus value at baseline.
Time Frame: Baseline to endpoint (6 weeks)
Population: All randomized participants with both baseline and post-baseline measures. Intention to Treat analysis.
Measure: Mean (Standard Deviation); unit: milligrams per deciliter
Arm/Group | Olanzapine | Placebo
Number analyzed (Participants) | 77 | 82
milligrams per deciliter
  Baseline | 91.81 (11.98) | 91.90 (10.13)
  Change from Baseline | 6.93 (23.72) | -0.55 (14.00)
Statistical Analysis 1: Comparison: Olanzapine vs Placebo; Test type: Superiority or Other; p = 0.007, ANOVA — P-value for Fasting Blood Glucose Change from Baseline; Type III sums of squares of ANOVA model: Ranked Change= Treatment + Pooled Investigator

10. Secondary Outcome: Clinically Significant Laboratory Values - Bilirubin Total Change From Baseline
Description: Change from baseline to endpoint in bilirubin total: Value of bilirubin total measure at endpoint minus value at baseline.
Time Frame: Baseline to endpoint (6 weeks)
Population: All randomized participants with both baseline and post-baseline measures. Intention to Treat analysis.
Measure: Mean (Standard Deviation); unit: micromoles per Liter
Arm/Group | Olanzapine | Placebo
Number analyzed (Participants) | 82 | 84
micromoles per Liter
  Baseline | 6.50 (3.46) | 6.65 (3.43)
  Change from Baseline | -1.56 (2.99) | -0.74 (3.03)
Statistical Analysis 1: Comparison: Olanzapine vs Placebo; Test type: Superiority or Other; p = 0.046, ANOVA — P-value for Bilirubin Total Change from Baseline; Type III sums of squares of ANOVA model: Ranked Change= Treatment + Pooled Investigator

11. Secondary Outcome: Clinically Significant Vital Signs - Body Mass Index Change From Baseline
Description: Change from baseline to endpoint in body mass index (an estimate of body fat derived by dividing body weight by height squared): Value of body mass index measure at endpoint minus value at baseline.
Time Frame: Baseline to endpoint (6 weeks)
Population: All randomized participants with both baseline and post-baseline measures. Intention to Treat analysis.
Measure: Least Squares Mean (Standard Error); unit: kilograms per square meters
Arm/Group | Olanzapine | Placebo
Number analyzed (Participants) | 100 | 101
kilograms per square meters | 1.18 (0.12) | 0.26 (0.12)
Statistical Analysis 1: Comparison: Olanzapine vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Type III sums of squares of ANCOVA model: Change= Treatment + Pooled Investigator + Baseline

12. Secondary Outcome: Clinically Significant Vital Signs - Weight Change From Baseline
Description: Change from baseline to endpoint: Value of weight measure at endpoint minus value at baseline.
Time Frame: Baseline to endpoint (6 weeks)
Population: All randomized participants with both baseline and post-baseline measures. Intention to Treat analysis.
Measure: Least Squares Mean (Standard Error); unit: kilograms
Arm/Group | Olanzapine | Placebo
Number analyzed (Participants) | 100 | 101
kilograms | 3.34 (0.34) | 0.70 (0.34)
Statistical Analysis 1: Comparison: Olanzapine vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Type III sums of squares of ANCOVA model: Change= Treatment + Pooled Investigator + Baseline

13. Secondary Outcome: Clinically Significant Vital Signs - Percentage of Participants With Baseline-to-Endpoint Weight Increase of at Least Seven Percent (7%)
Description: Percentages of participants in each group who experienced an increase in weight of at least 7% from baseline to endpoint.
Time Frame: Baseline to endpoint (6 weeks)
Population: All randomized participants with both baseline and post-baseline measures. Intention to Treat analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Olanzapine | Placebo
Number analyzed (Participants) | 100 | 101
percentage of participants | 22 | 3
Statistical Analysis 1: Comparison: Olanzapine vs Placebo; Test type: Superiority or Other; p < 0.001, Fisher Exact

ADVERSE EVENTS:
Groups:
- Olanzapine: Olanzapine: 15mg, capsules, PO at Q HS, daily for 1 week followed by 5-20mg, capsules, PO at Q HS daily for 5 weeks (6 weeks total). Divalproex: dose to maintain blood levels of 75-125 ug/mL, PO, BID, daily for 6 weeks (following d ose achieved in Study Period I)
- Placebo: Placebo: placebo capsules, PO, at Q HS, daily, for 6 weeks. Divalproex: dose to maintain blood levels of 75-125 ug/mL, PO, BID, daily for 6 weeks (following dose achieved in Study Period I).
Arm/Group | Olanzapine | Placebo
Serious Adverse Events (participants affected / at risk) | 3 | 5
Other Adverse Events (participants affected / at risk) | 80 | 63
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Olanzapine | Placebo
Asthenia (General disorders) | 0/101 (0) | 1/101 (1)
Chest pain (General disorders) | 0/101 (0) | 1/101 (1)
Death (General disorders) | 1/101 (1) | 0/101 (0)
Acute hepatic failure (Hepatobiliary disorders) | 1/101 (1) | 0/101 (0)
Head injury (Injury, poisoning and procedural complications) | 1/101 (1) | 0/101 (0)
Overdose (Injury, poisoning and procedural complications) | 0/101 (0) | 1/101 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1/101 (1) | 0/101 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0/101 (0) | 1/101 (1)
Hypoaesthesia (Nervous system disorders) | 0/101 (0) | 1/101 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0/101 (0) | 1/101 (1)
Bipolar I disorder (Psychiatric disorders) | 1/101 (1) | 1/101 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected / at risk (number of events):
Term (organ system) | Olanzapine | Placebo
Abdominal distension (Gastrointestinal disorders) | 3/101 (3) | 0/101 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1/101 (1) | 3/101 (3)
Dry mouth (Gastrointestinal disorders) | 13/101 (13) | 3/101 (3)
Dyspepsia (Gastrointestinal disorders) | 1/101 (1) | 3/101 (3)
Nausea (Gastrointestinal disorders) | 3/101 (3) | 1/101 (1)
Stomach discomfort (Gastrointestinal disorders) | 0/101 (0) | 3/101 (3)
Fatigue (General disorders) | 10/101 (12) | 4/101 (5)
Oedema peripheral (General disorders) | 6/101 (6) | 1/101 (2)
Nasopharyngitis (Infections and infestations) | 4/101 (4) | 7/101 (7)
Weight increased (Investigations) | 21/101 (21) | 4/101 (4)
Increased appetite (Metabolism and nutrition disorders) | 13/101 (13) | 5/101 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 3/101 (4) | 1/101 (1)
Akathisia (Nervous system disorders) | 3/101 (3) | 0/101 (0)
Dizziness (Nervous system disorders) | 3/101 (3) | 3/101 (4)
Headache (Nervous system disorders) | 5/101 (6) | 7/101 (7)
Sedation (Nervous system disorders) | 24/101 (25) | 4/101 (5)
Somnolence (Nervous system disorders) | 21/101 (23) | 6/101 (6)
Tremor (Nervous system disorders) | 9/101 (9) | 0/101 (0)
Agitation (Psychiatric disorders) | 2/101 (2) | 4/101 (4)
Insomnia (Psychiatric disorders) | 2/101 (2) | 6/101 (6)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0/101 (0) | 3/101 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 3/101 (3) | 0/101 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days